CLINICAL TRIAL: NCT00589446
Title: Investigation of Embryoscopy in Recurrent Pregnancy Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Collaborators: Herzliya Medical Center (Other)
Responsible Party: Prof. Howard Carp, MB, BS. FRCOG (Principal Investigator), Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SHEBA-05-3804-HC-CTIL
Record Dates: First submitted 2007-12-27; First posted 2008-01-09 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Recurrent Miscarriage
Keywords: Embryoscopy; recurrent miscarriage; missed abortion; Structural anomalies in recurrent miscarriage; Embryoscopically directed biopsy for karyotyping
MeSH Terms: conditions — Abortion, Habitual; Abortion, Missed | interventions — Hysteroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Embryoscopy will be evaluated in women with at least two previous miscarriages, after confirmation of missed abortion by ultrasound. Embryoscopy will only be performed in patients in whom curettage is clinically indicated, and will only be added to the D&C if there is a possibility of visualizing embryonic tissue, i:e. from approximately 5½ weeks onwards when there is an embryonic pole detected on ultrasound.
  Interventions: Device: Hysteroscope

INTERVENTIONS:
Device: Hysteroscope — An 8mm hysteroscope with irrigation channel and 30 degree view will be inserted into the uterus prior to curettage in cases of recurrent missed abortion

SUMMARY:
The purpose is to test the value of embryoscopy in women with missed abortions after recurrent miscarriages (at least two previous miscarriages) in the past. This project will assess two functions of embryoscopy:-

1. Whether embryoscopy allows the diagnosis of structural anomalies (disorganized embryos). This is a fetal cause of embryo loss which cannot be diagnosed by other means.
2. Whether embryoscopy allows an accurate biopsy of embryonic tissue for karyotyping.

However, it may be that embryoscopy will be found to have no advantage.

DETAILED DESCRIPTION:
In this project, embryoscopy will be evaluated in women with missed abortions (pregnancies which have ceased developing and in which the embryo is dead), after at least two previous (recurrent) miscarriages. The procedure will have two main purposes:- To allow the diagnosis of structural anomalies (disorganized embryos), and to allow an accurate biopsy of embryonic tissue for karyotyping. Hence, this procedure will lead to a more accurate diagnosis of the cause of recurrent miscarriage.

After confirmation of missed abortion by ultrasound, dilatation and curettage (D&C) is normally performed under general anesthetic to evacuate the uterus in missed abortions. In this project embryoscopy will be added to the standard D&C. An 8mm hysteroscope with irrigation channel and 300 view will be used with continuous saline flow. The embryo will be visualized, and the findings recorded. Biopsies will be taken for chromosomal analysis from the embryo and the placental villi. Embryoscopy will be performed with a hysteroscope which is in normal clinical use for investigating the uterine cavity, but for a slightly different indication.

The first stage will be a pilot study on 20 patients to judge the value of embryoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent miscarriage, (at least 2 consecutive miscarriages)
* Confirmation of missed abortion by ultrasound
* At least 5 1/2 weeks of gestation
* D & C is clinically indicated

Exclusion Criteria:

* Sporadic miscarriages
* Less than two consecutive miscarriages.
* If D & C is not clinically indicated

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2006-01; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To test the value of embryoscopy in women with missed abortions after recurrent miscarriages | Yearly

SECONDARY OUTCOMES:
Whether embryoscopy allows the diagnosis of structural anomalies | Annual
Whether embryoscopy allows an accurate biopsy of embryonic tissue for karyotyping. | Annual

CONTACTS AND LOCATIONS:
Overall Officials: Howard JA Carp, MB BS. FRCOG, Principal Investigator — Sheba Medical Center
Locations (2):
- Israel (2):
  - Herzlia Medical Center, Herzliya
  - Sheba Medical Center, Tel Litwinsky

REFERENCES:
- [Background] Philipp T, Philipp K, Reiner A, Beer F, Kalousek DK. Embryoscopic and cytogenetic analysis of 233 missed abortions: factors involved in the pathogenesis of developmental defects of early failed pregnancies. Hum Reprod. 2003 Aug;18(8):1724-32. doi: 10.1093/humrep/deg309. PMID 12871891
- [Result] Ferro J, Martinez MC, Lara C, Pellicer A, Remohi J, Serra V. Improved accuracy of hysteroembryoscopic biopsies for karyotyping early missed abortions. Fertil Steril. 2003 Nov;80(5):1260-4. doi: 10.1016/s0015-0282(03)02195-2. PMID 14607585
- [Result] Philipp T, Kalousek DK. Transcervical embryoscopy in missed abortion. J Assist Reprod Genet. 2001 May;18(5):285-90. doi: 10.1023/a:1016666301481. PMID 11464580